CLINICAL TRIAL: NCT00188201
Title: An Investigation of Cognitive Functioning and Brain Metabolites in Patients With Non-Cirrhotic Hepatitis-C Both Pre- and Post-Treatment With Antiviral Medication
Brief Title: Neurocognitive Functioning in Patients With Hepatitis C Pre- and Post-Treatment With Antiviral Medication
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: 01-0827-E; EOP-48307
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-11-29 (Estimated); Status verified 2005-09

CONDITIONS: Hepatitis C; Hepatitis B
Keywords: Hepatitis C; neucognitive functions; neuropsychological testing; antiviral treatment
MeSH Terms: conditions — Hepatitis C; Hepatitis B

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The estimated global prevalence of hepatitis C (HCV) infection is approximately 3% (170 million individuals). In Canada there are an estimated 240,000 people infected with HCV. The current study addresses the hypothesis that neurocognitive and neurochemical abnormalities may occur in individuals with HCV-infection who do not have liver cirrhosis or vasculitic neuropathy, and this may result from a direct effect of HCV on the Central Nervous System (CNS). The purpose of this study is to assess whether infection with the Hepatitis-C virus is associated with changes in thinking skills and brain chemistry, in patients who do not have liver cirrhosis. In addition, we are examining whether such changes in thinking skills and brain chemistry are reversed by antiviral treatment. We are also studying whether factors such as fatigue and depression have an effect on thinking skills in people with Hepatitis-C. In order to take into account the impact of having viral hepatitis, we will be comparing the results of the Hepatitis-C group to the results of a group of patients with Hepatitis-B, and to a group of individuals who do not have Hepatitis.

DETAILED DESCRIPTION:
The current proposal addresses the hypothesis that neurocognitive and neurochemical abnormalities may occur in individuals with HCV-infection who do not have liver cirrhosis or vasculitic neuropathy, and that this phenomenon may result from a direct effect of HCV on the Central Nervous System (CNS). Our hypothesis originated from the frequently reported complaints of forgetfulness and decreased ability to concentrate ('brain fog') in our patients with chronic HCV-infection, as well as from clinical observation of cognitive impairment in a moderate proportion of non-cirrhotic HCV-infected patients. Patients with HCV-infection also report significant impairment in most realms of everyday function, and greater reductions in quality of life (QOL) than individuals infected with the Hepatitis B virus (HBV). These results cannot be attributed to degree of liver inflammation, or the mode of acquisition of infection. Based on the well-established association between neurocognitive function and quality of life, it is reasonable to hypothesize that these QOL differences between HCV and HBV are the result of cerebral compromise in individuals infected with HCV, and consequent neuropsychiatric and neurocognitive dysfunction.

Non-cirrhotic HCV-infected patients were found to be impaired on speeded measures of sustained attention and working memory relative to control subjects. MRS results from the same study suggested that there may also be neurochemical changes associated with HCV that can be observed even in infected individuals with normal liver status (as determined by biopsy). In particular, an increase in choline ratios, was detected in the basal ganglia and white matter. This pattern appears to be specific to HCV-infection as abnormalities were not found in patients with Hepatitis-B infection. Furthermore, the degree of neurochemical abnormality was correlated with neuropsychological performance. Similar increases in choline levels have been reported in subcortical brain regions in individuals infected with HIV-1, even prior to the onset of symptomatic infection and signs of cognitive dysfunction.

Rationale: Mechanism through which HCV may have direct CNS effects A plausible mechanism for direct CNS effects of HCV involves passage of the virus into brain tissue through infection of circulating lymphocytes. In fact, a number of studies have revealed the presence of HCV RNA-negative strand (an intermediate of viral replication) within peripheral blood mononuclear cells (PMBC). However, the issue of extra-hepatic replication in PBMC remains controversial due to contrary findings and methodological criticisms. However, more recently Laskus and colleagues demonstrated the presence of HCV RNA-negative strand in PBMC in 40-60% of HCV-infected individuals with HIV-1 co-infection, and in a separate investigation determined the presence of HCV RNA-negative strand in monocytes/macrophages, CD4+ and CD8+ lymphocytes, and CD19+ cells in HCV/HIV-1 co-infected individuals. Thus, it is plausible that HCV enters the brain through circulating lymphocytes, and that consequent neuropsychiatric, neurocognitive, and neurochemical abnormalities are related to the presence of HCV in the CNS in a way that is not yet understood. Corroborating this hypothesis is the recent observation by Thomas and colleagues (personal communication) that HCV can be detected in the brain tissue of infected individuals upon neuropathological examination of autopsy tissue. This proposed mechanism for direct CNS effects of HCV-infection is similar to that which is thought to be the cause of HIV-1 associated neurocognitive impaiiment. Early in the course of the HIV-1 epidemic came the realization of frequent neurological complications, including neuropsychiatric, neurocognitive, and motor dysfunction. These symptoms could not be attributed to opportunistic infection of the CNS (e.g. toxoplasmosis; neoplasms), and often progressed to a stage of dementia, which came to be known as HIV-associated dementia (HAD). The incidence of HAD has declined drastically subsequent to the advent of antiretroviral treatment. HIV-1 is thought to enter the brain very early in the course of initial infection, possibly through the infection of peripheral monocytes and macrophages that cross the blood-brain barrier. In HAD, there is a complex and indirect mechanism of CNS damage that may occur years after initial HIV-1 infection, usually under conditions of immunocompromise. HIV-1 does not directly infect neurons, but rather replicates within brain macrophages and microglia. These cells subsequently become immunoactive, and release secretory neurotoxic substances that ultimately lead to a breakdown of homeostatic mechanisms, and a consequent cascade of inflammatory events. The resulting metabolic encephalopathy damages, and eventually destroys CNS neurons. The most prominent neuropathological features of HAD occur in white matter and deep grey matter regions of the brain, and include myelin pallor, multinucleated giant cells, and occasionally encephalitis characterized by disseminated, multifocal microgranulomas composed of elongated microglia, macrophages, and lymphocytes. Thus, given preliminary findings of extra-hepatic replication within PBMC as a plausible mechanism for infiltration of CNS by HCV-infected lymphocytes, neuropathological detection of HCV within the CNS, clinical observation and patient complaints of cognitive deficits, and reduction in HRQOL beyond that observed in chronic HBV-infection, it is possible that HCV may have direct CNS effects that elicit a consequent inflammatory reaction that interferes with neuronal function in a manner similar to the neuropathological processes associated with HIV-1 infection. Furthermore, there are parallels between MRS findings for HIV-1 and those reported in HCV-infection in non-cirrhotic patients. In particular, HIV-1 is marked by an increase in choline-containing compounds (Cho), similar to the preliminary findings of Forton and colleagues (1999; 2000). This increase in subcortical Cho can be found in HIV-1 positive patients even in the absence of cognitive dysfunction, suggesting it may be a very early marker of CNS involvement. Other changes, notably a decrease in N-acetylaspartate, are apparent in HIV-1 infected individuals with significant neuropsychological impairment, indicating an evolution of CNS disease. Of importance, antiretroviral therapy appears to reverse the Cho abnormalities, and also results in significant improvements in neurocognitive function.

Objectives Phase I In the first phase, we will determine whether non-cirrhotic individuals with chronic HCV-infection (who do not have cryoglobulinemia) manifest abnormalities in brain biochemistry and neurocognitive performance. This will be accomplished by comparing HCV-infected individuals to subjects with HBV-infection (to control for the effects of viral hepatitis), and to an age-matched control group on measures of neurocognitive performance and MRS after careful screening to rule out the presence of other conditions that may affect cognitive performance. We will also determine whether there is a relationship between MRS-quantified brain biochemistry and neurocognitive performance. Finally, we will reveal the determinants of neurocognitive impairment and neurochemical abnormalities using multivariate analyses, to evaluate the relative contribution of other clinical parameters associated with HCV-infection, such as fatigue, mood / psychiatric symptoms, serum aminotransferase levels, degree of fibrosis, viral load.

Phase II In the second phase of our investigation, we will determine whether HCV-infected patients who achieve a sustained virological response to antiviral therapy (no HCV RNA detectable in serum) will show amelioration of cerebral metabolite abnormalities and cognitive impairment at follow-up (6 months following the cessation of treatment), compared to patients who do not respond to antiviral treatment and compared to an age-matched control group (the same control subjects tested in Phase I of the investigation). In the group that does not respond to treatment, MRS abnormalities will remain unchanged, or may worsen. A control group is particularly important for the NP assessment aspect of the investigation, in order to account for practice effects that may result from repeated administration of NP tests. Patients with HBV-infection will not be re-tested at this point, because we do not expect to see any abnormalities in this group at the initial assessment point. In addition, if HBV-infected patients were started on antiviral treatment following their liver biopsy, it is likely that they will still be receiving treatment 1-5 years later. The rationale for timing the final assessment of HCV patients 6 months after the cessation of antiviral therapy involves the known neuropsychiatric sequelae of treatment with Interferon (which may otherwise affect the cognitive assessment). Efficacy of antiviral treatment of HCV with Interferon and ribavirin At the time of this submission, treatment with IFNa2b plus ribavirin is the standard of care for patients with chronic HCV-infection. However, recently published data indicates that when interferon is pegylated (covalently bound to polyethylene glycol), efficacy is markedly enhanced in comparison to standard IFNa2b plus ribavirin. Enhanced efficacy is likely due to the sustained elevation of IFN in serum, due to delay of its renal excretion. Thus, weekly (rather than three times weekly) injections are required. Pilot study data indicates that the efficacy of pegylated IFN alfa-2a plus ribavirin is even more effective. This portion of the investigation is an add-on to a safety study involving treatment with 6 or 12 months of Pegylated Interferon alfa-2a plus ribabvirin (UHN # 01-0082). We expect that the rate of sustained virological responders in non-cirrhotic patients will be approximately 54%.

METHODS: Subjects - In total, 150 subjects will participate in the investigation, 100 of which will be assessed on two different occasions, approximately 1.5 years apart. Fifty patients with chronic Hepatitis C infection (HCV), fifty with chronic Hepatitis B infection (HBV), and fifty healthy control subjects will be recruited to participate in the investigation. All participants will undergo screening procedures to rule out conditions that can affect cognitive function. Those that are deemed eligible on the basis of the inclusion and exclusion criteria will participate in the first phase of the investigation in which they will be assessed with Physical, Neurological, Psychiatric, and Neuropsychological examinations, as well as with Magnetic Resonance Spectroscopy. In the second phase of the investigation, HCV patients and control subjects will be reassessed after an interval of 1.0 to 1.5 years to determine whether antiviral treatment is effective at ameliorating neurocognitive and brain biochemical abnormalities identified in the first phase of the investigation.

Materials: Assessments and Procedures Screening Assessments Liver Biopsy All HCV and BBV patients who have received a liver biopsy as part of their clinical management will be eligible to participate in the current investigation, although no patient will receive a biopsy for the purposes of this investigation. Instead, participants will be recruited from the pool of subjects who are receiving clinical care at the UHNTWH Liver Clinic who have had a recent liver biopsy performed, and will be progressing to treatment (both HBV and HCV patients).

Laboratory Assessment HCV and HBV patients will undergo a screening laboratory assessment that will consist of hematological assessment, blood chemistry, and urinalysis as per the protocol for the clinical trial that this investigation is being added on to (UHN # 01-0082). In addition, supplementary laboratory assessments will be conducted to screen for other parameters that may be related to cognitive function. In particular, the following tests will be performed: RBC/Folate, Hb Urea, Electrolytes, Bl2, TSH, Cryoglobulins, INR, Albumin.

Physical Evaluation All HCV and HBV patients will be assessed by the Principle Investigator for clinical signs of liver disease, and will also have a general physical examination as specified in the clinical trial protocol (UHN # 01-0082). HBV patients will be assessed by the Principle Investigator in a similar manner. The results of this assessment will be used to screen for signs of clinically significant liver disease (e.g. stigmata, asterixis, liver size, spleen size, jaundice, ascites or edema, as well as for other conditions related to liver disease that could possibly affect cognition and thus exclude the participant from participation in the investigation (e.g. cryogloubulinemia).

Neurological Examination: Patients will be examined by the study neurologist for the presence of conditions that would result in exclusion from the investigation. The neurologist will also examine the patients for signs of peripheral neuropathy that could indicate the presence of cryoglobulinemia (e.g. dysesthesia or hypesthesia, motor weakness, exaggerated deep tendon reflexes, and positive pyramidal signs). In addition, the neurological examination will be conducted during the final visit in order to determine whether any of the neurological side effects known to be associated with Interferon therapy have persisted beyond the 6 month wash-out period.

Psychiatric Examination: The patient will be examined by the study psychiatrist to determine current and lifetime presence of psychiatric diagnoses that could result in their exclusion from the investigation. Of specific concern are psychiatric diagnoses that could have an impact on cognitive function (e.g. Major Depression, Bipolar Disorder, Substance Abuse disorder, Antisocial Personality Disorder).

ELIGIBILITY:
Inclusion Criteria:

* patients attending Liver Clinic at Toronto Western Hospital, Toronto, ON, Canada
* Fluent in English
* Men and women between the ages of 18 and 65
* Subjects must provide written informed consent to participate
* Control subjects: negative for both HBV, HCV, and HIV

Additional Inclusion Criteria For HCV and HBV patients:

* patient is a candidate for antiviral treatment
* non-cirrhotic as determined by recent liver biopsy (<2 years prior to assessment)
* HCV subjects: positive for HCV RNA, negative for HBV and HIV
* HBV subjects: positive for HBV RNA and negative for HCV and HIV

Exclusion Criteria:

presence of any of the following medical conditions:

* Thyroid dysfunction, or other endocrine disorder
* Major psychiatric disease, especially major depression and bipolar disorder
* Vitamin B12 or folate deficiency
* Unstable cardiovascular disease (especially atrial fibrillation)
* Unstable diabetes
* Haemophilia (depending on frequency of medication usage)
* The presence of other viral infections (HIV; syphilis)
* Use of pharmaceuticals known to affect cognitive function
* Current alcohol use greater than 2 units per day, or prior history of alcoholism
* Use of illicit drugs within 2 years, or prior prolonged history
* History of intravenous drug use within the past 5 years
* History of any of the following neurological conditions: head injury with loss of consciousness greater than 30min., history of stroke, dementia, seizure disorder,recent substance abuse disorder (within 2 years), learning disability
* Postmenopausal and perimenopausal female participants, unless hormone replacement therapy has been administered consistently for 2 years (on the basis that they may have concentration and memory dysfunction related to cholinergic deficits)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: E.J.L (Jenny) Heathcote, MD, Principal Investigator — UHN - Toronto Western Hospital, University of Toronto
Locations (1):
- Liver Clinic, Toronto Western Hospital, UHN., Toronto, Ontario, Canada